CLINICAL TRIAL: NCT07021703
Title: A Open-label, Randomized Study to Evaluate the Safety and Tolerability of Freeze-dried Human Rabies Vaccine (Human Diploid Cells) Administered to Participants With Different Immunization Schedules
Brief Title: A Clinical Trial of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIM2301-Ⅰ-01
Record Dates: First submitted 2025-05-15; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): The Participants received 1 dose of AIM2301 on day 0, 3, 7, 14 and 28, a total of 5 doses
  Interventions: Biological: Freeze-dried Human Rabies Vaccine（Human Diploid Cell）, Essen
- Group2 (Experimental): The Participants received 2 dose of AIM2301 on day 0, 1 dose of AIM2301 on day7 and 21, a total of 4 doses
  Interventions: Biological: Freeze-dried Human Rabies Vaccine（Human Diploid Cell），Zagreb

INTERVENTIONS:
Biological: Freeze-dried Human Rabies Vaccine（Human Diploid Cell）, Essen — This vaccine is produced by Ningbo Rongyu Biological Pharmaceutical Co., Ltd.. Participants will receive AIM2301 by intramuscular injection.
  Receive on the day 0, 3, 7, 14 and 28, a total of 5 doses
  Other Names: AIM2301
  Arms: Group1
Biological: Freeze-dried Human Rabies Vaccine（Human Diploid Cell），Zagreb — This vaccine is produced by Ningbo Rongyu Biological Pharmaceutical Co., Ltd.. Participants will receive AIM2301 by intramuscular injection.
  Receive 2 doses on day 0, 1 dose on day 7 and day 21, a total of 4 doses.
  Other Names: AIM2301
  Arms: Group2

SUMMARY:
The Phase 1 clinical trial of the freeze-dried human rabies vaccine (human diploid cells) will be conducted on participants aged 10 to 60. This study will design a single-arm, randomized, open-access trial with different immunization schedules (5-dose schedule and 2-1-1 schedule) to evaluate the safety and tolerability of the vaccine in participants aged 10 to 60

DETAILED DESCRIPTION:
This trial will adopt a single-arm, randomized, open-label experimental design, with a planned enrollment of 60 participants, comprising 30 individuals aged 10-17 years and 30 aged 18-60 years. Initially, 30 participants in the 18-60 age group will be enrolled and randomly assigned in a 1:1 ratio to either the 5-dose schedule group or the 2-1-1 schedule group. Participants in the 5-dose schedule group will receive five doses of the trial vaccine according to the immunization schedule of days 0, 3, 7, 14, and 28. Those in the 2-1-1 schedule group will receive four doses of the trial vaccine according to the immunization schedule of day 0 (two doses), day 7, and day 21. Following the administration of the first dose, safety will be monitored for 7 days among participants aged 18-60 years. If no criteria for trial suspension/termination are met, an additional 30 participants in the 10-17 age group will be enrolled and randomly assigned in a 1:1 ratio to either the 5-dose schedule group or the 2-1-1 schedule group, following the same immunization schedules as described above.

Adverse events (AEs) that occur from the first dose of vaccination through 30 days post-completion of the full vaccination regimen will be collected. Serious adverse events (SAEs), pregnancy-related events (including pregnancy outcomes, delivery characteristics, neonatal conditions, and growth and development within one month postpartum for female participants), reported from the first dose of vaccination through 6 months post-completion of the full vaccination regimen, will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* (1) The participants' ages range from 10 to 60 years old (≥10 years old and <61 years old).

  (2) Participants aged 10 to 17 and their guardians can provide valid identification documents, and participants aged 18 to 60 can provide their own valid identification documents.

  (3) Participants aged 10 to 17 and their guardians, as well as participants aged 18 to 60, can sign the informed consent form voluntarily to participate in the trial, fully understand the trial procedures, the risks of participating in the trial, and other intervention measures that can be chosen if they do not participate in the trial, etc.

  (4) Possess basic reading and writing skills, and be capable of reading, understanding and filling in diary cards and contact cards; (5) Female participants with fertility must also meet the following conditions: 1) They have taken effective contraceptive measures within two weeks prior to participating in this trial; 2) Have no plans to have children within 6 months from the start of participating in this trial until the full vaccination. 3) Understand and agree to take effective contraceptive measures during the trial period (from the first dose to within 6 months after the full vaccination). Effective contraceptive measures include: condoms (for men), intrauterine devices, oral contraceptives (excluding emergency contraceptives), sterilization, abstention, injection or implantable contraception, sustained-release local contraceptives, hormone patches, diaphragms, cervical caps, etc. External ejaculation and safe period contraception are not regarded as effective contraceptive measures.

Exclusion Criteria:

* For the standards marked with *, if the participants have the circumstances stipulated in the standard, the visit can be rescheduled when they no longer have these circumstances

  1. After inquiry, it is found that there is a history of rabies vaccination or the use of passive immunization preparations for rabies virus.
  2. There was a history of injury from rabies virus-susceptible animals (such as cats and dogs) before the first dose of vaccination;
  3. The axillary body temperature of the participants on the day of enrollment was ≥37.3℃*;
  4. Those whose various examination results during the screening period are abnormal and are determined by clinicians to be of clinical significance;
  5. Women who have a positive urine pregnancy test before vaccination (on the day of vaccination), or who, after assessment, cannot rule out the possibility of pregnancy or are breastfeeding;
  6. Hypertension that cannot be controlled by medication, such as systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg for participants aged 18 years and above before enrollment;
  7. Allergy to any component of the vaccine used in the test, such as human albumin, sucrose, or maltose;
  8. Those with a history of severe allergies in the past, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, local allergic necrosis reaction (Arthus reaction), severe urticaria, allergic bronchitis, acquired angioedema, etc.
  9. Has been diagnosed with congenital or acquired immune system diseases Such as Human Immunodeficiency Virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease or other immune diseases that researchers determine may affect the evaluation of the trial;
  10. Known or suspected of having serious diseases, including severe respiratory diseases, liver and kidney diseases, cardiovascular and cerebrovascular diseases, malignant tumors, and other chronic diseases that are poorly controlled, etc.
  11. Abnormal coagulation function (such as deficiency of coagulation factors, coagulation disorders, abnormal platelets) or coagulation disorders diagnosed by a doctor;
  12. Anplenia or functional anplenia, as well as anplenia or splenectomy caused by any circumstances;
  13. Previous or current clearly diagnosed neurological or mental disorders (including but not limited to dementia, schizophrenia, bipolar disorder, etc.) or confirmed epilepsy, convulsions, as well as other neurological or mental disorders that the researcher deems unsuitable for participation in this trial;
  14. It is planned to receive such treatment within 30 days after the first dose of vaccination and the full course of vaccination, such as long-term systemic glucocorticoid therapy (used continuously for 2 weeks or more, at a dose of 2mg/kg/ day or 20mg/ day prednisone or an equivalent dose); Local medications (such as ointments, eye drops, inhalants or nasal sprays) are allowed;
  15. Have received or plan to receive immunoenhancers or inhibitors, immunoglobulins or blood-related products throughout the trial period within 3 months prior to enrollment;
  16. Have received attenuated live vaccines within 14 days before enrollment, and subunit vaccines or inactivated vaccines within 7 days *;
  17. Within 3 days before enrollment, have suffered from acute diseases or be in the acute attack stage of chronic diseases *;
  18. Antipyretic, analgesic and antihistamine drugs were used within 3 days before enrollment.
  19. Currently participating in or planning to participate in other clinical trials during this clinical trial;
  20. According to the researcher's judgment, due to various medical, psychological, social conditions or other circumstances contrary to the trial protocol, or the participants' inability to comply with the requirements of the trial protocol.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of AE and AR within 30 minutes after each dose of vaccination | within 30 minutes after each dose of vaccination
  After each dose of the investigational vaccine is administered, participants should be observed on-site for 30 minutes. The contents of safety observation include any medical events occurring in participants.
  The severity and relevance of AEs shall be determined in accordance with the guidance for adverse event grading criteria and the guidance for relevance determination.
The occurrence of AE and AR within 7 days after each dose of vaccination | within 7 days after each dose of vaccination
  After each dose of vaccine is administered, a Diary Card will be issued to participants. Participants and/or their guardians should measure body temperature daily from Day 0 to Day 7 and observe/record all adverse events (AEs) as well as concomitant medications/vaccines according to the requirements of the Diary Card.
  The severity and relevance of AEs shall be determined in accordance with the guidance for adverse event grading criteria and the guidance for relevance determination.
The occurrence of AE and AR within 30 days from the first dose of vaccination to the full course of vaccination | within 30 days from the first dose of vaccination to the full course of vaccination
  Solicited and unsolicited adverse events from the first dose vaccination to 30 days after full-course vaccination shall be collected through diary cards and contact cards.
  The severity and relevance of AEs shall be determined in accordance with the guidance for adverse event grading criteria and the guidance for relevance determination.
Abnormal changes /Occurrence of clinically significant abnormal changes in laboratory test indicators | the third day after the first dose of vaccination
  Abnormal changes /Occurrence of clinically significant abnormal changes in laboratory test indicators (blood biochemistry, blood routine and urine routine) on the third day after the first dose of vaccination
The occurrence of serious adverse events | within 6 months from the first dose of vaccination to the full course of vaccination.
  The occurrence of serious adverse events within 6 months from the first dose of vaccination to the full course of vaccination.
  SAE assessed include any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No